CLINICAL TRIAL: NCT07401225
Title: Transcranial Magnetic Stimulation as Treatment for Persistent PTSD in Texas Youth
Brief Title: TMS for PTSD in Youth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Texas Child Mental Health Care Consortium: TCMHCC (Unknown)
Responsible Party: Principal Investigator, Amy Garrett, PhD, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002052; NECMHR02 (Other: Texas Childhood Mental Healthcare Consortium (TCMHCC))
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Posttraumatic Stress Disorder in Adolescents
Keywords: Transcranial Magnetic Stimulation; Non-invasive treatment; Mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Open label single group design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- TMS treatment group (Experimental): Each treatment visit will take about 1.5 hours. Participants will receive up to 4 TMS treatment sessions during the visit, with each session lasting about 10-minutes. After the TMS sessions, there will be a brief visit with a psychotherapist.
  Interventions: Device: MagPro R30 with robotic arm

INTERVENTIONS:
Device: MagPro R30 with robotic arm — TMS will be delivered to the right anterior dorsolateral frontal cortex. The accelerated protocol consists of 1,800 TMS pulses per session, delivered at intensity ranges designed to deliver depth-corrected E-fields of 80-95 volts/meter. The exact intensity will be determined when the participant's treatment plan is developed. Once a patient's TMS treatment plan has been created, it will be used for every treatment session for that participant.

SUMMARY:
The purpose of this study is to test whether transcranial magnetic stimulation, or TMS, is an acceptable and helpful treatment for ongoing symptoms of posttraumatic stress syndrome disorder (PTSD) in 12-20 year olds. Ongoing PTSD refers to symptoms that continue after completing trauma-focused psychotherapy. About 1 in 4 patients need additional help to overcome PTSD after completing psychotherapy. Currently, scientists do not know the best way to help adolescents with persistent PTSD, and this study will test TMS as a possible treatment, and hopefully lead to future studies including more people.

DETAILED DESCRIPTION:
Trauma is a common occurrence among youth. Almost 60% of American youths experience a traumatic event before age 18, such as physical or sexual abuse, sudden loss of caregivers, or witnessing violence in the community or the home. Distress after a significantly traumatic event is to be expected, but for some youths, symptoms of posttraumatic stress disorder (PTSD) linger for months or years, and can become chronic if left untreated. Symptoms of PTSD can include upsetting memories, avoidance of reminders, and emotional numbing, and other symptoms. These symptoms can create difficulties for family relationships, friendships, and schoolwork. Currently, the most effective treatment for PTSD is talk therapy (trauma-focused psychotherapy). However, sometimes young people continue to have symptoms of PTSD after completing talk therapy, and it is currently not known the best way to help with these persistent symptoms.

In this study, the total length of time participants will be involved in the study is about 16-weeks. During that time, participants will be asked to attend approximately 6 research visits and 10 treatment visits, for a total of 16 visits. The 6 research visits include a screening visit, an interview visit, 2 MRI visits, and 2 follow-up visits. The screening, interview, and follow-up visits can be completed virtually, over zoom. The study will include 2 MRI visits and 10 treatment visits. Virtual follow-up visits will be conducted 1 and 3 months after completion of treatment and will include interviews and questionnaires about participants symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females; Age 12-20
2. Have previously completed at least 9 sessions of trauma-focused therapy in our clinical trial or in the community
3. Have current self-reported symptom score of 20 or greater on the UCLA PTSD Reaction index
4. Willing to attend 10 TMS treatment sessions within a 30-day period
5. Fluent in English

Exclusion Criteria:

1. History of seizures
2. History of head injury with loss of consciousness and concussive sequelae
3. Brain abnormality such as tumor or other observable abnormality
4. Currently receiving psychotherapy or TMS treatment
5. Currently pregnant
6. MRI contraindications (metal in body, orthodontic braces)
7. Diagnosis of bipolar 1 or a psychotic disorder

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Side Effects of TMS treatment | Day 1 of treatment through Day 30
  number of side effects reported per participant
Number of Adverse Events | Day 1 of treatment through Day 30
  Number of adverse events experienced by study participants through the treatment phase of the study
Completion rate of Treatment | Day 1 of treatment through Day 30
  Number of participants that completed the TMS treatment

SECONDARY OUTCOMES:
Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5)(CAPS-5) | Baseline to 90 days
  The CAPS-5 score range for total symptom severity is 0 to 80, calculated by summing the severity ratings (0-4) for 20 PTSD symptoms, with higher scores indicating greater severity; scores below 31-33 often suggest subclinical or non-diagnostic levels, while scores above this range can indicate probable PTSD.
Assessment of Depression using Patient Health Questionnaire-9 (PHQ-9) | Baseline to Day 30
  Patients rate 9 common depressive symptoms (e.g., feeling down, trouble sleeping, low energy, poor appetite, concentration issues, feeling bad about self, restlessness/slowed down, thoughts of being better off dead/hurting self).
  Scoring: Each symptom gets 0-3 points, totaling 0-27. A lower score indicates less depression.

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Garrett, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- UT Health Department of Psychiatry, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
requests for data will be considered on a case-by-case basis